CLINICAL TRIAL: NCT05292508
Title: Rapid Diagnostic Testing for C-reactive Protein to Differentiate Bacterial and Viral Infection in Febrile Patients to Reduce Antimicrobial Use in Remote Health Care Centers of Gulmi District of Nepal: a Cluster Randomized Controlled Trial
Brief Title: Comparison of Rates of Antimicrobial Use in Febrile Patients With or Without the Use of C-reactive Protein Blood Test
Acronym: CREATIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Patan Academy of Health Sciences (Other)
Collaborators: Gulmidarbar Rural Municipality (Unknown); Dhurkot Rural Municipality (Unknown); Resunga Municipality (Unknown)
Responsible Party: Principal Investigator, Amit Arjyal, Assistant Professor, Patan Academy of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1-2022
Record Dates: First submitted 2022-02-23; First posted 2022-03-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Acute Febrile Illness; Use of Antimicrobial Agents; C-reactive Protein Level
Keywords: C-Reactive Protein; Acute Febrile Illness; Viral Infection; Bacterial Infection; Antimicrobial Drug; CRP Rapid Test
MeSH Terms: conditions — Virus Diseases; Bacterial Infections

STUDY DESIGN:
Intervention Model Description: We will conduct a Cluster Randomized Controlled Trial (cRCT) at eight Health Posts of Gulmi District. Eight Health Posts will be randomly allocated to the intervention arm (use of rapid diagnostic test for C-reactive protein) and the other will be allocated to the control arm. Thus, there will be four Health Posts each in the intervention and control arms.
Who Masked: Outcomes Assessor
Masking Description: A study investigator will make the assessment of outcome for each patient after reviewing the patients electronic clinical records. This electronic record will not have information about the health post where the trial recruitment took place. The allocation arm will also not be disclosed in this record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRP Tests in addition to Usual Standard of Care (Experimental): For the clusters (health posts) in this arm, the health worker will prick the finger of the eligible patient using a lancet device following aseptic precautions. A very small drop (10 microliters) of whole blood will be obtained which will be added to specimen dilution buffer and the dipstick will be placed into the diluted sample. It will be removed after the liquid rises and the timer will be started and result will be interpreted in 5 minutes. Interpretation of CRP levels: Only red color line (No blue line): <10 mg/L One blue line: 10-40 mg/L Two blue lines: 40-80 mg/L Three blue lines: >80 mg/L. CRP levels of 40 mg/L or above will be considered as increased CRP levels. The decision on antimicrobial use and other treatments will be made with the help of CRP results in addition to information obtained from the history and physical examination.
  Interventions: Diagnostic Test: C-reactive Protein Rapid Diagnostic Test
- Usual Standard of Care Alone (No Intervention): For the clusters (health posts) in this control arm, Usual Standard of Care Alone will be provided. This usual standard of care is given to patients with febrile illness at health posts. Commonly, this involves taking a brief history and conducting a simple physical examination followed by symptomatic treatment such as paracetamol, cough medication or analgesics such as NSAIDs. Often antimicrobial treatment is also prescribed based on clinical suspicion of bacterial infection.

INTERVENTIONS:
Diagnostic Test: C-reactive Protein Rapid Diagnostic Test — In the intervention arm in addition to Usual Standard of Care, CRP Testing will be performed. In this test, health worker at health post will prick the finger of the patient using a lancet device following aseptic precautions. A very small drop (10 microliters) of whole blood will be obtained. This will be added to specimen dilution buffer. Then the sample will be mixed by inverting the tube upside down 10-15 times. Then the yellow dip area of the dipstick will be placed into the diluted sample. It will be held there until the liquid rises to the result area by capillary action. The the dipstick is removed from the solution and placed in a horizontal position. The timer will be started and result will be interpreted in 5 minutes. Treatment decision making regarding the use of antimicrobials will be conducted with the help of CRP test results and other clinical features.
  Arms: CRP Tests in addition to Usual Standard of Care

SUMMARY:
In Health Posts of rural areas operated by the Government of Nepal, there are limitations of tests to differentiate between bacterial and viral infections. Due to this, health workers are obliged to prescribe antimicrobials (antibacterials) just on the basis of clinical features. This can lead to irrational use of antimicrobials, consequently contributing to antimicrobial resistance. C-reactive protein is the marker of inflammation which rises during bacterial infection but rarely rises during viral infection. The investigators wish to compare the effect on antimicrobial usage of using CRP(C-Reactive Protein) test, a rapid diagnostic test used to differentiate bacterial and viral infection, with usual standard of care, by carrying out a cluster-randomized controlled trial. The investigators plan to carry out this study in eight Health Posts of Resunga, Dhurkot and Gulmi-Durbar Municipalities of Gulmi District. The investigators will randomly allocate four Health Posts (clusters) to the intervention arm- CRP TESTS in addition to Usual Standard of Care, and four Health Posts (clusters) to the control arm- Usual Standard of Care Alone. The investigators plan to study all patients above one year of age presenting with fever or a history of reported fever with a duration of up to 7 days in Health Posts. Primarily, the investigators will assess the rates of antimicrobial use per patient who presents with febrile illness. Secondarily, the investigators will also assess the outcome of illness of the patient such as need for subsequent hospital admission or severe or complicated illness. This testing method will supplement the existing methods to differentiate bacterial and viral infections based on history and clinical examination by health professionals as a part of usual standard of care in the Health Posts included in this study.

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines antimicrobial resistance (AMR) as a situation where drugs used to treat microbial infection caused by bacteria, viruses, fungi and parasites no longer work to treat infection because of the changes in these microbes over time. Though this process of development of AMR is a natural process, it is accelerated by the overuse and misuse of antimicrobials (Mladenovic-Antic et al, 2016, pp.532-537). There were an estimated 1.27 million deaths attributable to bacterial AMR globally in 2019 (Murray et al, 2022). It is estimated that in India every year around sixty thousand newborns die due to AMR (Laxminarayan et al, 2013, pp.1057-1098). As big as the death toll due to AMR is, the economic costs are also significant. Even in a setting of a developed country like the US, direct healthcare cost of AMR is over 6 billion US dollars (CDC, 2019). Nepal is one of the developing countries of the world located in South Asia between India and China. AMR is an increasing problem in Nepal and some of the most common causes for it are excessive use of antimicrobials in animal husbandry and unnecessary use of antimicrobials for treatment of febrile illness (Rijal et al, 2021, pp. 1-14; Acharya and Wilson, 2021, p.105). Currently, bacteria like Escherichia coli, Klebsiella pneumoniae, Streptococcus pneumoniae, Shigella spp., Vibrio cholera, Neisseria gonorrheae and Staphylococcus aureus are increasingly resistant to the most first-line and some second-line antimicrobials (Acharya and Wilson, 2021 p.105; Basnyat et al, 2015, pp.102-111). Thus antimicrobial resistance (AMR) presents a great threat to public health.

Nepal has its own National Antibiotic Treatment Guideline and according to this even the smallest government healthcare units like health posts can prescribe antimicrobials. These health posts lack microbiology laboratory access and the health worker has to prescribe antimicrobials based upon their history and examination findings which may lead to unnecessary prescription of antimicrobials against viral illness. This challenge of unavailability of laboratory tests can be tackled by introducing point-of-care rapid diagnostic test to detect C-reactive protein to differentiate between bacterial and viral infections. C-reactive protein is the marker of inflammation which rises in blood during bacterial infection but rarely rises during viral infection (Phommasone et al, 2015, pp.1-6). This method has already been used in other developing countries like Laos, Thailand, Myanmar, Malaysia and Vietnam, which have similar socio-economic conditions like that of Nepal (Phommasone et al, 2015, pp.1-6; Althaus et al, 2019, pp.e119-e131; Lubell et al, 2018, pp.1-6; Haenssgen et al, 2018, pp.1-12). Antimicrobials are rarely prescribed based on an absolute certainty of a bacterial infection. The use of point-of-care rapid diagnostic test offers an easy, affordable and a working solution to this problem and helps in judicial use of antimicrobials (O'Neill, 2016). Although it is known that CRP testing can differentiate bacterial and viral infections, the extent to which it can reduce antimicrobial use in a rural health-post setting of Nepal and thus play a role in limiting the emergence of antimicrobial resistance is not known. If this study shows significant reduction in antimicrobial prescription without any adverse clinical outcome, the test kit can be implemented nationally in all low resource health care settings in Nepal.

ELIGIBILITY:
Inclusion Criteria:

* History of reported fever or fever greater than 100.4◦F (38◦C) with duration of illness up to 7 days
* Duration of fever less than or equal to 7 days
* Can connect with mobile phone for follow up

Exclusion Criteria:

* Child younger than 1 year
* Main complaint being trauma or injury
* Symptoms requiring hospital referral
* Impaired consciousness
* Inability to take oral medication
* Convulsions
* Confirmed malaria
* Confirmed urinary tract infection
* Local skin infection
* Dental abscess or infection
* Suspicion of tuberculosis
* Any symptom other than fever present for more than 14 days
* Any bleeding such as from skin, nose and gums.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 924 (Estimated)
Dates: Start 2023-02-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Use of antimicrobial | On the 1 day of recruitment to the study
  The investigators will record if the patient was prescribed antimicrobial at the time of presenting to the health post during the current acute febrile illness. This outcome will be recorded as Yes/No

SECONDARY OUTCOMES:
Complicated Illness | One month from recuitment
  The investigators will record this as outcome of disease after contacting the patient at one month of recruitment and ask whether the patient developed any complications or not. This outcome will be recorded as Complicated Illness (Yes/No). Complicated illness will be defined as need for prolonged course of treatment for more than one week, need to change the initial treatment provided at the health post and give rescue treatment, any severe illness or death. This outcome will be recorded as Yes/No
Referral to hospital | One month from recruitment
  The investigators will record this outcome after contacting the patient at one month of recruitment and ask whether the patient was referred to a hospital. This outcome will be recorded as Yes/No
Admission to hospital | One month from recuitment
  The investigators will record this outcome after contacting the patient at one month of recruitment and ask whether the patient was admitted to hospital. This outcome will be recorded as Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Amit Arjyal, MBBS, DPhil, Principal Investigator — Patan Academy of Health Sciences
Locations (1):
- Paralmi Health Post, Resunga Nagarpalika, Lumbini, Nepal

IPD SHARING:
Plan to Share IPD: No